CLINICAL TRIAL: NCT00006042
Title: Non-Myeloablative Allogeneic Bone Marrow Transplantation for Hematologic Malignancies Using Haploidentical Donors: A Phase I Trial of Pre-Transplant Cyclophosphamide
Brief Title: Cyclophosphamide Plus Bone Marrow Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068057, J9966; P30CA006973 (NIH); JHOC-J9966; JHOC-99110501; NCI-G00-1816
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent adult Hodgkin lymphoma; Burkitt lymphoma; refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent/refractory childhood Hodgkin lymphoma; stage II adult lymphoblastic lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Hodgkin Disease; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Filgrastim; Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of cyclophosphamide plus bone marrow transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the minimum effective dose of pretransplant cyclophosphamide to induce engraftment of haploidentical allogeneic bone marrow without the use of myeloablative conditioning in patients with hematologic malignancies.
* Determine the incidence and severity of graft versus host disease and nonhematologic toxicities with this treatment regimen in these patients.
* Correlate the pretreatment phenotypic and functional immunologic characteristics in these patients in relation to risk of graft rejection with this treatment regimen.

OUTLINE: This is a dose-escalation study of cyclophosphamide.

Patients receive fludarabine IV over 1 hour on days -6 to -2; cyclophosphamide IV over 1 hour on days -6, -5, and 3; total body irradiation on day -1; and allogeneic bone marrow transplantation on day 0. Patients also receive tacrolimus IV or orally twice a day on days 4-50; oral mycophenolate mofetil on days 4-35; and filgrastim (G-CSF) subcutaneously or IV starting on day 4 and continuing until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of cyclophosphamide until the minimum effective dose necessary to induce chimerism without unacceptable toxicity in these patients is determined.

Patients are followed at 2 and 6 months, at one year, and then annually thereafter.

PROJECTED ACCRUAL: At least 23 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with any of the following diagnoses:

  * Chronic myelogenous leukemia

    * Chronic phase 1

      * Failed prior interferon alfa therapy OR
      * Relapsed after prior autologous stem cell transplantation
    * Chronic phase 2
  * Acute leukemia

    * Standard risk

      * Age over 60 years
      * Complete remission 1 (CR1)
    * High risk

      * High WBC at presentation, unfavorable cytogenetics, mixed lineage, delayed response to induction chemotherapy
      * CR1
      * Complete remission 2 or higher
  * Acute lymphocytic leukemia

    * CR1 or higher
  * Myelodysplastic syndrome

    * Untreated OR
    * CR1
  * Acute myeloid leukemia in CR1
  * Chronic lymphocytic leukemia

    * Rai stage III or IV OR
    * Received prior autologous stem cell transplantation
  * Multiple myeloma

    * Stage II or III
    * Stable or progressive disease after prior chemotherapy OR
    * Received prior autologous stem cell transplantation
  * Non-Hodgkin's Lymphoma
  * Hodgkin's lymphoma
* Ineligible for or refused autologous or standard allogeneic bone marrow transplantation
* Ineligible for bone marrow transplantation from an HLA matched, sibling donor or from an HLA matched, unrelated donor
* Must have an HLA mismatched, related donor (3-5 out of 6)

PATIENT CHARACTERISTICS:

Age:

* 0.5 to 70

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 3.1 mg/dL

Renal:

* Not specified

Cardiovascular:

* Left ventricular ejection fraction at least 35%

Pulmonary:

* FEV_1 and FVC at least 40% of predicted OR
* FEV_1 and FVC at least 60% in patients who have received prior thoracic or mantle radiotherapy

Other:

* HIV negative
* No other debilitating medical or psychiatric illness that would preclude study compliance
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior transfusions from donor

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim J. Fuchs, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] O'Donnell PV, Luznik L, Jones RJ, Vogelsang GB, Leffell MS, Phelps M, Rhubart P, Cowan K, Piantados S, Fuchs EJ. Nonmyeloablative bone marrow transplantation from partially HLA-mismatched related donors using posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2002;8(7):377-86. doi: 10.1053/bbmt.2002.v8.pm12171484.